CLINICAL TRIAL: NCT01092702
Title: A Pilot Study of Varenicline for Tobacco Dependence Treatment in Recovering Alcoholic Smokers: the Clinical Trial
Brief Title: Varenicline For Smokers In Recovery From Alcohol Dependence
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: James Taylor Hays, MD, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-00672
Record Dates: First submitted 2010-03-19; First posted 2010-03-25 (Estimated); Results first posted 2010-11-30 (Estimated); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Tobacco Abstinence
Keywords: Tobacco Dependence; Smoking; Tobacco Cessation
MeSH Terms: conditions — Tobacco Use Disorder; Smoking; Tobacco Use Cessation | interventions — Varenicline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Varenicline (Other): Everyone on study will receive Varenicline daily for 12 weeks
  Interventions: Drug: Varenicline

INTERVENTIONS:
Drug: Varenicline — During the first week varenicline will be started at a dose of 0.5 mg once daily for days 1-3; then 0.5 mg twice daily for days 4-7. Target quit date is set at day 8. Varenicline is then continued for weeks 2-12 at a dose of 1 mg twice daily.
  Other Names: Varenicline Tartrate; Chantix (in the USA); Champix (in Europe)

SUMMARY:
The goal of this proposal is to explore the potential effectiveness of varenicline to treat tobacco dependence among recovering alcoholic smokers who, as a group, are at high risk for tobacco-caused morbidity and mortality. In this open-label phase II clinical trial, we are proposing to enroll 32 recovering alcoholic smokers who are motivated to stop smoking. After the initial up titration of varenicline in week 1, all 32 subjects will receive a total of 2 mg/day of varenicline for 12 weeks. In addition to receiving varenicline, all subjects will receive brief behavioral counseling and our standard intervention at each visit during participation in the study.

DETAILED DESCRIPTION:
This is an open-label, phase II clinical trial. All subjects will be screened for study eligibility after providing informed consent. During the clinic screen visit the subjects are informed of the study, the study informed consent is signed by the subject and staff member, a series of screening tests are conducted and screening criteria are reviewed. Once enrolled in study, the subject will return for a face to face clinic visit weekly for the first 4 weeks (visits 3-6) and then biweekly for the last 8 weeks(visits 7-10). Target quit day is the day after visit 3 (week 1 visit).

During the first week varenicline will be started at a dose of 0.5 mg once daily for days 1-3; then 0.5 mg twice daily for days 4-7. Target quit date is set at day 8. Varenicline is then continued for weeks 2-12 at a dose of 1 mg twice daily.

Subjects will return weekly for 4 weeks then bi-weekly for the remaining 8 weeks. The study end-date will be Week 12, which is also the end-of-treatment date.

ELIGIBILITY:
Inclusion Criteria:

1. Male or non-pregnant female cigarette smoker; 18-years-of-age or older and reporting smoking at least an average of 10 cigarettes per day for the past year.
2. A history of alcohol dependence based on DSM IV criteria as assessed by the Alcohol Dependence Scale and the physician investigator
3. A minimum of 6 months of abstinence from alcohol use as assessed by the physician investigator
4. Subject must be able to complete all the study visits
5. Subject must be in general good health as determined by medical history, physical exam and physician investigator
6. Subject must provide written informed consent to participate in the study.

Exclusion Criteria:

1. Current treatment with another investigational drug.
2. Current use (within past 30 days) of nicotine replacement therapy, bupropion, rimonabant, varenicline, nortriptyline, clonidine, or other medications known to be effective for treating tobacco dependence.
3. Subject has current (past 30 days) major depressive disorder or has a history of another psychiatric disorder such as psychosis or bipolar disorder.
4. Current (past 6 months) drug abuse corroborated by the Drug Abuse Screening Test (DAST-20) and physician interview.
5. Regular use of other tobacco products (i.e. pipe, cigar, smokeless tobacco) within the past 30 days.
6. Females who are pregnant, lactating or likely to become pregnant during the trial and not willing to use an acceptable form of contraception during the medication phase. For women of child-bearing potential, a pregnancy test will be performed prior to entry into the study and at the end of the medication phase.
7. A history of a major cardio-vascular event in the past 3 months including unstable angina, acute MI or coronary angioplasty.
8. Known allergy to varenicline.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2008-04; Primary Completion 2008-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James T Hays, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Nicotine Research Program, Rochester, Minnesota, United States

REFERENCES:
- [Result] Hays JT, Croghan IT, Schroeder DR, Ebbert JO, Hurt RD. Varenicline for tobacco dependence treatment in recovering alcohol-dependent smokers: an open-label pilot study. J Subst Abuse Treat. 2011 Jan;40(1):102-7. doi: 10.1016/j.jsat.2010.08.009. Epub 2010 Oct 13. PMID 20947286

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began on 04/14/2008 and finished on 08/28/2008. Recruitment was in the general community of Rochester, Minnesota
Pre-assignment Details: All potential participants consenting to enrollment completed a series of screening questionnaires. The questionnaires included demographic information, alcohol and smoking history, the the Center for Epidemiological Studies-Depressed Mood Scale, DAST-20, medical history and physical exam.
Groups:
- Varenicline: Everyone on study received Varenicline (2 mg/day) daily for 12 weeks
Period: Overall Study
Arm/Group | Varenicline
Started | 32
Completed | 23
Not Completed | 9
Not completed — Withdrawal by Subject | 7
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Arm/Group | Varenicline
Number analyzed (Participants) | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 32
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.9 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 22
Region of Enrollment [Number; unit: participants]
  United States | 32
cigarettes per day [Mean (Standard Deviation); unit: cigarettes per day] — Self reported average number of cigarettes smoked per day over the preceding 6 months prior to study enrollment.
  cigarettes per day | 20.3 (5.0)
Duration of alcohol recovery [Median (Full Range); unit: months] — Self reported number of months in recovery from alcohol dependence prior to study enrollment.
  months | 29 [6 to 217]

OUTCOME MEASURES:

1. Primary Outcome: Biochemically Confirmed Abstinence From Smoking
Description: The primary endpoint of this trial is biochemically confirmed 7-day point prevalence smoking abstinence at the end of the medication phase (week 12). Self-reported abstinence from smoking (not even a puff) over the last 7-days will be considered biochemically confirmed by an expired air CO of <8 ppm. Subjects who discontinue the study or have a missed visit for any reason will be classified as smoking for that visit.
Time Frame: 12 weeks from start of medication
Measure: Number; unit: participants
Arm/Group | Varenicline
Number analyzed (Participants) | 32
participants | 10

ADVERSE EVENTS:
Time Frame: Adverse Events were collected for the 12 weeks of study medication phase.
Arm/Group | Varenicline
Serious Adverse Events (participants affected / at risk) | 0/32
Other Adverse Events (participants affected / at risk) | 18/32
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Varenicline (N=32)
Nausea (Gastrointestinal disorders) | 9
Sleep Disturbance (General disorders) | 6
Abnormal Dreams (General disorders) | 5
Depression/Anxiety (Psychiatric disorders) | 5
other gastrointestinal (Gastrointestinal disorders) | 3
behavior Change (Psychiatric disorders) | 2
Headache (General disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes